CLINICAL TRIAL: NCT01287572
Title: Efficiency of Ventilation During Conscious Sedation of Pediatric Patients Undergoing Minor Procedures in the Pediatric Intensive Care Unit
Brief Title: Efficiency of Ventilation During Conscious Sedation in the Pediatric Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Prof. Yakov Sivan, Tel-Aviv Sourasky Medical Center
Other Study IDs: TASMC-10-YS-319-CTIL
Record Dates: First submitted 2011-01-24; First posted 2011-02-01 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Conscious Sedation
Keywords: TcCO2; sedation; procedure; PICU

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Conscious sedation group: Pediatric patients 0 to 18 years requiring conscious sedation for procedures done in the pediatric ICU excluding burned patients or patients with severe eczema or other skin disease.

SUMMARY:
Pediatric patients admitted to the intensive care unit and requiring conscious sedation for minor surgical procedures are at risk to hypoventilate and retain CO2.

The rise in CO2 levels is not well described and unpredicted. In this study the investigators will monitor CO2 levels transcutaneously using SDMS (SenTec digital Monitoring System) a device recently approved for clinical use. The hypothesis is ventilation of patients undergoing conscious sedation is compromised and CO2 levels might rise significantly to levels that potentially can effect hemodynamics.

In order to avoid hemodynamic changes proper and routine monitoring is recommended.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patirnts 0- 18 years admitted to the pediatric intensive care unit
* patients requiring minor surgical procedures (e.g. bronchoscopy, central venous line placement, lumbar puncture, intracranial pressure monitoring device insertion)

Exclusion Criteria:

* skin disease
* burns to thorax

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric patirnts 0- 18 years admitted to the pediatric intensive care unit and undergoing minor procedures
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-02 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
TcCO2 level | One year
  Transcutaneous measurement of patients undergoing conscious sedation

CONTACTS AND LOCATIONS:
Overall Officials: Yakov Sivan, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center; Efraim Sadot, MD, Study Director — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel